CLINICAL TRIAL: NCT04587232
Title: Adaptation and Validation of the Mini Osteoarthritis Knee and Hip Quality of Life (Mini-OAKHQoL) Questionnaire in Turkish Population
Brief Title: Turkish Version of Mini Osteoarthritis Knee and Hip Quality of Life Questionnaire
Acronym: Mini-OAKHQoL
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2017.493
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Knee Osteoarthritis; Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Turkish version of Mini Osteoarthritis Knee and Hip Quality of Life Questionnaire — Turkish version of Mini Osteoarthritis Knee and Hip Quality of Life Questionnaire (Mini-OAKHQoL) was derived from the Turkish version of OAKHQoL questionnaire, which was developed to assess the quality of life (QoL) in subjects with lower limb osteoarthritis. It includes five subscales: physical activities, mental health, pain, social support, social functioning; with three additional independent items addressing sexual life, professional life, and fear of being dependent. The numerical rating scales in the items range from 0 (worst) to 10 (best). Scores were obtained by computing the means of the item scores in each subscale. The last three items' score (independent items) becomes the corresponding score.
Diagnostic Test: Nottingham Health Profile — Standardized questionnaire to investigate the health-related quality of life. NHP is a general is used to measure health problems perceived by the patient. It comprises 6 sections. The sum of the items within each section ranges from 0 to 100, and the total score ranges from 0 to 600. The higher score shows a worse quality of life.
Diagnostic Test: Short form 36 — Standardized questionnaire to investigate the general health-related quality of life. The SF-36 questionnaire is a generic quality of life questionnaire and consists of 8 subscales, with 36 items. The scores ranges from 0 to 100 and the high score indicates good health.
Diagnostic Test: Western Ontario and McMaster — Standardized questionnaire to investigate the health status of patients with osteoarthritis. The WOMAC OA index assesses the symptomatic severity and disability with pain, stiffness, and physical function domains. Each subscale was summated to a maximum score of 20, 8, and 68, respectively, with the higher scores corresponding worst health status.

SUMMARY:
In this paper, the adaptation of the Mini-OAKHQoL questionnaire in the Turkish population analyzing the feasibility, reliability, and validity of the questionnaire was documented.

DETAILED DESCRIPTION:
Knee and hip osteoarthritis are common diseases that play an important role in health-related quality of life (HR-QoL). Assessing HR-QoL with a disease- and site-specific HR-QoL is more advantageous than generic scales. In that concept, to our knowledge, there is not any osteoarthritis- and lower limb-specific HR-QoL instrument to use in Turkey. Mini-OAKHQoL was derived from the OAKHQoL questionnaire, which was developed to assess the quality of life (QoL) in subjects with lower limb osteoarthritis. Its good psychometric properties have recently been shown and validation studies have been done in several populations. Mini-OAKHQoL's validation study has not been done before in Turkey. The aim is to investigate the validity and reliability of the Turkish version of the Mini-OAKHQoL. Patients diagnosed with knee or hip osteoarthritis were recruited. For cross-cultural adaptation, items of Mini-OAKHQoL were selected from the interrelated Turkish version of the OAKHQoL study in which the adaptation process had already done. Missing data, floor effect, and ceiling effect were calculated. Reliability analysis with internal consistency and test-retest reliability were discovered. Face, content, convergent, and divergent validities were applied.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic knee or hip OA
* between 18-75 years

Exclusion Criteria:

* history of inflammatory disease,
* a disease involving cognitive deficit and psychiatric illness,
* knee or hip surgery within one year,
* another disease of the lower limbs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with uni-or bilateral symptomatic knee or hip OA from the Rheumatology Division of Physical Medicine and Rehabilitation Department, Marmara University Faculty of Medicine, with the age between 18-75 years were included.
Sampling Method: Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2017-10-14 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Turkish version of Mini Osteoarthritis Knee and Hip Quality of Life Questionnaire (Mini-OAKHQoL) | 0 day
  Turkish version of Mini Osteoarthritis Knee and Hip Quality of Life Questionnaire (Mini-OAKHQoL) was derived from the Turkish version of OAKHQoL questionnaire, which was developed to assess the quality of life (QoL) in subjects with lower limb osteoarthritis. It includes five subscales: physical activities, mental health, pain, social support, social functioning; with three additional independent items addressing sexual life, professional life, and fear of being dependent. It asks for the impact of the knee or hip OA on their QoL over the last month while filling the items. The numerical rating scales in the items range from 0 (worst) to 10 (best). Scores were obtained by computing the means of the item scores in each subscale. The social support and social functioning subscales are questioned inverse but scored similarly to the "0 (worst)-10 (best) concept. The last three items' score (independent items) becomes the corresponding score.

SECONDARY OUTCOMES:
test-retest reliability | 14 days
  For test-retest reliability, participants were asked to refill the Turkish version of Mini Osteoarthritis Knee and Hip Quality of Life Questionnaire after two weeks from the initial assessment.
internal consistency | 0 day
  The reliability of the Turkish version of Mini Osteoarthritis Knee and Hip Quality of Life Questionnaire was assessed by internal consistency using Cronbach's alpha coefficient and test-retest reliability using intraclass correlation coefficients.
correlations for construct validity | 0 day
  Convergent and divergent validities were analyzed to determine the construct validity. Convergent validity was assessed by correlating the Turkish version of Mini Osteoarthritis Knee and Hip Quality of Life (Mini-OAKHQoL) questionnaire score with the subsets of Nottingham Health Profile (NHP), Short form 36 (SF-36), and Western Ontario and McMaster questionnaire (WOMAC). The correlations of the Mini-OAKHQoL with parameters that are not directly related to the health-related quality of life, such as age, body mass index, and disease duration were assessed for divergent validity.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Tuncay Duruöz, Professor, Study Director — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Guillemin F, Rat AC, Goetz C, Spitz E, Pouchot J, Coste J. The Mini-OAKHQOL for knee and hip osteoarthritis quality of life was obtained following recent shortening guidelines. J Clin Epidemiol. 2016 Jan;69:70-8. doi: 10.1016/j.jclinepi.2015.06.010. Epub 2015 Jun 22. PMID 26111768
- [Background] Gonzalez Saenz de Tejada M, Bilbao A, Herrera C, Garcia L, Sarasqueta C, Escobar A. Validation of the Mini-OAKHQOL for use in patients with osteoarthritis in Spain. Clin Rheumatol. 2017 Aug;36(8):1855-1864. doi: 10.1007/s10067-017-3611-z. Epub 2017 Mar 28. PMID 28353088